CLINICAL TRIAL: NCT05926661
Title: Support Tool for Families of High-Risk Children With Heart Disease During Hospital Admission and After Discharge
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per NIH guidelines study does not meet criteria for clinical trial
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Deepika Thacker, Pediatric Cardiologist, Nemours Children's Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Support Tools; U54GM104941-10 (NIH)
Record Dates: First submitted 2023-05-30; First posted 2023-07-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Heart Disease Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent/Caregiver of high-risk children with heart disease (Other): The parent/caregivers of high-risk children with heart disease coming to the Nemours Cardiac Center for care will be offered a "support tool" and will be asked for it's acceptance and feasibility through their experience.
  Interventions: Other: NCC Support Toolkit

INTERVENTIONS:
Other: NCC Support Toolkit — Pre-discharge intervention-
  * Set expectations for parents/caregivers to spend time bedside and attend rounds
  * iPad for the families to use the Nemours App, download education materials and Facetime communication with medical personnel.
  * Download Nemours App and teach them how to use it
  * Education materials- to ease the use of medications, Oxygen and feeding
  * Assistance with transportation, child care, parental work schedule for discharge teaching
  Post Discharge intervention (Day 1-2):
  • Video/Facetime call with the family to check equipment, home environment and answer questions about medications and formula
  Post discharge intervention (Day 3-7):
  • Phone call to the family to ensure transportation for their first follow-up appointment, answer questions about medications, Oxygen and feeding.

SUMMARY:
The goal of this study is to pilot the "support tool" in the Nemours Cardiac Center to assess acceptability and feasibility. This tool will be offered to 5 high-risk families, and they will be asked to complete a survey. In addition, healthcare providers including bed-side nurses and cardiologists will be asked to complete a survey to assess the feasibility of the tool.

DETAILED DESCRIPTION:
Despite advances in the care of children with heart disease, those affected often remain in need of complex care after hospital discharge. Multiple medications, tube feeds, and medical equipment are a few of the care needs parents face upon leaving the hospital. Unsurprisingly, many parents report problems in the transition of care from the hospital to the home. Clinical providers express frustration related to challenges with family education and communication around the time of discharge. Research is required to identify intervention strategies to improve parent/ caregiver confidence with caring for their child after discharge and reduce unintended resource utilization after discharge including clinical deterioration, unplanned 30-day readmissions, emergency department (ED) visits and nonadherence to outpatient appointments.

In Aim 1 of the study, the investigators identified the modifiable barriers, perceived needs, and opportunities for intervention to support parents/ caregivers in meeting the care needs of the high-risk child with heart disease after discharge by conducting semi-structured qualitative interviews with parents/ caregivers and healthcare personnel. And based on participants' responses, the investigators developed a support tool to improve parent/ caregiver comfort with caring for the high-risk child and improve post discharge outcomes. The objective of this study is to pilot this support tool in 5 high-risk families in Nemours Cardiac Center and assess the acceptability and feasibility based on their experience.

ELIGIBILITY:
Parent/Caregiver Group-

Inclusion Criteria:

• Parents of a child with congenital heart disease and planned discharge from the Nemours Cardiac Center.

Exclusion Criteria:

• Non-English and Non-Spanish speaking families.

The Healthcare providers group is pre-identified and they will be invited to provide feedback through semi-structured qualitative interviews only. They will not receive any intervention. Their participation will be voluntary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of support tool | 12 weeks
  By administering surveys to 5 families
Feasibility of support tool | 12 weeks
  By administering surveys to the bed-side nurses and cardiologists.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Thacker, MD, Principal Investigator — Nemours Children's Hospital
Locations (1):
- Nemours Children's Hospital, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahle WT, Spray TL, Wernovsky G, Gaynor JW, Clark BJ 3rd. Survival after reconstructive surgery for hypoplastic left heart syndrome: A 15-year experience from a single institution. Circulation. 2000 Nov 7;102(19 Suppl 3):III136-41. doi: 10.1161/01.cir.102.suppl_3.iii-136. PMID 11082376
- [Background] Jacobs JP, Quintessenza JA, Burke RP, Bleiweis MS, Byrne BJ, Ceithaml EL, Decampli WM, Giroud JM, Perryman RA, Rosenkranz ER, Wolff G, Posner V, Steverson S, Blanchard WB, Schiebler GL. Analysis of regional congenital cardiac surgical outcomes in Florida using the Society of Thoracic Surgeons Congenital Heart Surgery Database. Cardiol Young. 2009 Aug;19(4):360-9. doi: 10.1017/S1047951109990151. Epub 2009 Jul 6. PMID 19575843
- [Background] Harlan GA, Nkoy FL, Srivastava R, Lattin G, Wolfe D, Mundorff MB, Colling D, Valdez A, Lange S, Atkinson SD, Cook LJ, Maloney CG. Improving transitions of care at hospital discharge--implications for pediatric hospitalists and primary care providers. J Healthc Qual. 2010 Sep-Oct;32(5):51-60. doi: 10.1111/j.1945-1474.2010.00105.x. Epub 2010 Jul 23. PMID 20854359
- [Background] Co JP, Ferris TG, Marino BL, Homer CJ, Perrin JM. Are hospital characteristics associated with parental views of pediatric inpatient care quality? Pediatrics. 2003 Feb;111(2):308-14. doi: 10.1542/peds.111.2.308. PMID 12563056
- [Background] Freed GL, Uren RL. Hospitalists in children's hospitals: What we know now and what we need to know. J Pediatr. 2006 Mar;148(3):296-9. doi: 10.1016/j.jpeds.2005.12.048. No abstract available. PMID 16615954
- [Background] Connor JA, Kline NE, Mott S, Harris SK, Jenkins KJ. The meaning of cost for families of children with congenital heart disease. J Pediatr Health Care. 2010 Sep-Oct;24(5):318-25. doi: 10.1016/j.pedhc.2009.09.002. Epub 2010 Jan 6. PMID 20804952
- [Background] Faraoni D, Nasr VG, DiNardo JA. Overall Hospital Cost Estimates in Children with Congenital Heart Disease: Analysis of the 2012 Kid's Inpatient Database. Pediatr Cardiol. 2016 Jan;37(1):37-43. doi: 10.1007/s00246-015-1235-0. Epub 2015 Jul 17. PMID 26184611
- [Background] Demianczyk AC, Behere SP, Thacker D, Noeder M, Delaplane EA, Pizarro C, Sood E. Social Risk Factors Impact Hospital Readmission and Outpatient Appointment Adherence for Children with Congenital Heart Disease. J Pediatr. 2019 Feb;205:35-40.e1. doi: 10.1016/j.jpeds.2018.09.038. Epub 2018 Oct 23. PMID 30366772
- [Background] Fixler DE, Pastor P, Sigman E, Eifler CW. Ethnicity and socioeconomic status: impact on the diagnosis of congenital heart disease. J Am Coll Cardiol. 1993 Jun;21(7):1722-6. doi: 10.1016/0735-1097(93)90393-f. PMID 8496543
- [Background] Nembhard WN, Salemi JL, Ethen MK, Fixler DE, Dimaggio A, Canfield MA. Racial/Ethnic disparities in risk of early childhood mortality among children with congenital heart defects. Pediatrics. 2011 May;127(5):e1128-38. doi: 10.1542/peds.2010-2702. Epub 2011 Apr 18. PMID 21502234
- [Background] DiMatteo MR, Haskard KB, Williams SL. Health beliefs, disease severity, and patient adherence: a meta-analysis. Med Care. 2007 Jun;45(6):521-8. doi: 10.1097/MLR.0b013e318032937e. PMID 17515779
- [Background] Islam S, Yasui Y, Kaul P, Mackie AS. Hospital Readmission of Patients With Congenital Heart Disease in Canada. Can J Cardiol. 2016 Aug;32(8):987.e7-987.e14. doi: 10.1016/j.cjca.2015.12.018. Epub 2015 Dec 29. PMID 26968390
- [Background] Mackie AS, Ionescu-Ittu R, Pilote L, Rahme E, Marelli AJ. Hospital readmissions in children with congenital heart disease: a population-based study. Am Heart J. 2008 Mar;155(3):577-84. doi: 10.1016/j.ahj.2007.11.003. PMID 18294499
- [Background] Kogon B, Jain A, Oster M, Woodall K, Kanter K, Kirshbom P. Risk factors associated with readmission after pediatric cardiothoracic surgery. Ann Thorac Surg. 2012 Sep;94(3):865-73. doi: 10.1016/j.athoracsur.2012.04.025. Epub 2012 Jun 8. PMID 22682942
- [Background] Saharan S, Legg AT, Armsby LB, Zubair MM, Reed RD, Langley SM. Causes of readmission after operation for congenital heart disease. Ann Thorac Surg. 2014 Nov;98(5):1667-73. doi: 10.1016/j.athoracsur.2014.05.043. Epub 2014 Aug 15. PMID 25130076
- [Background] Knowles RL, Bull C, Wren C, Dezateux C. Mortality with congenital heart defects in England and Wales, 1959-2009: exploring technological change through period and birth cohort analysis. Arch Dis Child. 2012 Oct;97(10):861-5. doi: 10.1136/archdischild-2012-301662. Epub 2012 Jun 29. PMID 22753769
- [Background] Zheng G, Wu J, Chen P, Hu Y, Zhang H, Wang J, Zeng H, Li X, Sun Y, Xu G, Wen S, Cen J, Chen J, Guo Y, Zhuang J. Characteristics of in-hospital mortality of congenital heart disease (CHD) after surgical treatment in children from 2005 to 2017: a single-center experience. BMC Pediatr. 2021 Nov 23;21(1):521. doi: 10.1186/s12887-021-02935-2. PMID 34814864
- [Background] Pasquali SK, Jacobs ML, He X, Shah SS, Peterson ED, Hall M, Gaynor JW, Hill KD, Mayer JE, Jacobs JP, Li JS. Variation in congenital heart surgery costs across hospitals. Pediatrics. 2014 Mar;133(3):e553-60. doi: 10.1542/peds.2013-2870. Epub 2014 Feb 24. PMID 24567024
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Forster AJ, Clark HD, Menard A, Dupuis N, Chernish R, Chandok N, Khan A, van Walraven C. Adverse events among medical patients after discharge from hospital. CMAJ. 2004 Feb 3;170(3):345-9. PMID 14757670
- [Background] Moore C, Wisnivesky J, Williams S, McGinn T. Medical errors related to discontinuity of care from an inpatient to an outpatient setting. J Gen Intern Med. 2003 Aug;18(8):646-51. doi: 10.1046/j.1525-1497.2003.20722.x. PMID 12911647
- [Background] Hansen LO, Young RS, Hinami K, Leung A, Williams MV. Interventions to reduce 30-day rehospitalization: a systematic review. Ann Intern Med. 2011 Oct 18;155(8):520-8. doi: 10.7326/0003-4819-155-8-201110180-00008. PMID 22007045
- [Background] Tong HJ, Qiu F, Fan L. Effect of hospital discharge plan for children with type 1 diabetes on discharge readiness, discharge education quality, and blood glucose control. World J Clin Cases. 2021 Feb 6;9(4):774-783. doi: 10.12998/wjcc.v9.i4.774. PMID 33585623
- [Background] Parikh K, Hall M, Kenyon CC, Teufel RJ 2nd, Mussman GM, Montalbano A, Gold J, Antoon JW, Subramony A, Mittal V, Morse RB, Wilson KM, Shah SS. Impact of Discharge Components on Readmission Rates for Children Hospitalized with Asthma. J Pediatr. 2018 Apr;195:175-181.e2. doi: 10.1016/j.jpeds.2017.11.062. Epub 2018 Feb 1. PMID 29395170
- [Background] Mockenhaupt R, Woodrum A. Developing evidence for structural approaches to build a culture of health: a perspective from the Robert Wood Johnson Foundation. Health Educ Behav. 2015 Apr;42(1 Suppl):15S-19S. doi: 10.1177/1090198115575100. PMID 25829114
- [Background] Fortune K, Becerra-Posada F, Buss P, Galvao LAC, Contreras A, Murphy M, Rogger C, Keahon GE, de Francisco A. Health promotion and the agenda for sustainable development, WHO Region of the Americas. Bull World Health Organ. 2018 Sep 1;96(9):621-626. doi: 10.2471/BLT.17.204404. Epub 2018 Jul 27. PMID 30262943
- [Background] Weiss ME, Sawin KJ, Gralton K, Johnson N, Klingbeil C, Lerret S, Malin S, Yakusheva O, Schiffman R. Discharge Teaching, Readiness for Discharge, and Post-discharge Outcomes in Parents of Hospitalized Children. J Pediatr Nurs. 2017 May-Jun;34:58-64. doi: 10.1016/j.pedn.2016.12.021. Epub 2017 Jan 10. PMID 28087088
- [Background] Gottlieb LM, Garcia K, Wing H, Manchanda R. Clinical interventions addressing nonmedical health determinants in Medicaid managed care. Am J Manag Care. 2016 May;22(5):370-6. PMID 27266438
- [Background] Czajkowski SM, Powell LH, Adler N, Naar-King S, Reynolds KD, Hunter CM, Laraia B, Olster DH, Perna FM, Peterson JC, Epel E, Boyington JE, Charlson ME. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015 Oct;34(10):971-82. doi: 10.1037/hea0000161. Epub 2015 Feb 2. PMID 25642841
- [Background] Sood E, Karpyn A, Demianczyk AC, Ryan J, Delaplane EA, Neely T, Frazier AH, Kazak AE. Mothers and Fathers Experience Stress of Congenital Heart Disease Differently: Recommendations for Pediatric Critical Care. Pediatr Crit Care Med. 2018 Jul;19(7):626-634. doi: 10.1097/PCC.0000000000001528. PMID 29533356
- [Background] Hennink MM, Kaiser BN, Marconi VC. Code Saturation Versus Meaning Saturation: How Many Interviews Are Enough? Qual Health Res. 2017 Mar;27(4):591-608. doi: 10.1177/1049732316665344. Epub 2016 Sep 26. PMID 27670770
- [Background] Hennink MM, Kaiser BN, Weber MB. What Influences Saturation? Estimating Sample Sizes in Focus Group Research. Qual Health Res. 2019 Aug;29(10):1483-1496. doi: 10.1177/1049732318821692. Epub 2019 Jan 10. PMID 30628545
- [Background] Varaei S, Vaismoradi M, Jasper M, Faghihzadeh S. Iranian nurses self-perception -- factors influencing nursing image. J Nurs Manag. 2012 May;20(4):551-60. doi: 10.1111/j.1365-2834.2012.01397.x. Epub 2012 Feb 27. PMID 22591156
- [Background] Draucker CB, Martsolf DS, Ross R, Rusk TB. Theoretical sampling and category development in grounded theory. Qual Health Res. 2007 Oct;17(8):1137-48. doi: 10.1177/1049732307308450. PMID 17928484
- [Background] Beck CT. Grounded theory: overview and application in pediatric nursing. Issues Compr Pediatr Nurs. 1996 Jan-Mar;19(1):1-15. doi: 10.3109/01460869609026851. PMID 8920496
- [Background] Shoemaker SJ, Wolf MS, Brach C. Development of the Patient Education Materials Assessment Tool (PEMAT): a new measure of understandability and actionability for print and audiovisual patient information. Patient Educ Couns. 2014 Sep;96(3):395-403. doi: 10.1016/j.pec.2014.05.027. Epub 2014 Jun 12. PMID 24973195
- [Background] Vaismoradi MJ, J; Turunen, H; Snelgrove, S. Theme development in qualitative content analysis and thematic analysis. Journal of Nursing Education and Practice. 2016;6:100-110.

DOCUMENTS (1):
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT05926661/ICF_000.pdf